CLINICAL TRIAL: NCT06805565
Title: A Phase IIa, Randomized, Double-blind, Placebo Controlled, Parallel Group, Multi-center Trial to Evaluate the Efficacy and Safety of ONO-1110 in Patients With Social Anxiety Disorder
Brief Title: A Study of ONO-1110 in Patients With Social Anxiety Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-1110-08; jRCT2031240578 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Social Anxiety Disorder (SAD)
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-1110 (Experimental)
  Interventions: Drug: ONO-1110; Drug: Placebo
- Placeo (Placebo Comparator)
  Interventions: Drug: ONO-1110; Drug: Placebo

INTERVENTIONS:
Drug: ONO-1110 — ONO-1110 tablets once a day
Drug: Placebo — Placebo tablets once daily

SUMMARY:
To Evaluate the Efficacy and Safety of ONO-1110 in Patients with Social Anxiety Disorder

ELIGIBILITY:
Inclusion Criteria:

1. Japanese participants (sex not specified)
2. Participants who, in the opinion of the principal (or sub-investigator), are capable of understanding the content of the clinical trial and complying with its requirements
3. Participants diagnosed with social anxiety disorder based on DSM-5-TR (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision) criteria, as determined through an interview using the M.I.N.I. (Mini-international neuropsychiatric interview)
4. Outpatients
5. Participants with a LSAS-J (Liebowitz Social Anxiety Scale Japanese version) total score of 70 or higher and a CGI-S (Clinical global impression-Severity) score of 4 or higher

Exclusion Criteria:

1. Participants with a current or past history of psychiatric or neurological disorders that meet any of the following criteria:

   * Participants with a comorbid psychiatric disorder other than social anxiety disorder as defined by DSM-5-TR (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision) (assessed using the M.I.N.I. (Mini-international neuropsychiatric interview))
   * Participants with a comorbid or past history of schizophrenia or other psychotic disorders as defined by DSM-5-TR (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision)
   * Participants with neurodevelopmental disorders, neurocognitive disorders, or personality disorders (excluding avoidant personality disorder) as defined by DSM-5-TR
2. Participants who have been primarily diagnosed with a disorder other than social anxiety disorder according to DSM-5-TR (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision) criteria within 24 weeks prior to screening
3. Participants with a MADRS (Montgomery Åsberg Depression Rating Scale) total score of 15 or higher
4. Participants who, in the opinion of the principal (or sub-investigator), have not responded to at least two different SSRIs (Selective serotonin reuptake inhibitor), each administered at an adequate dose for at least 10 weeks, in treating social anxiety disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in L-SAS J(Liebowitz Social Anxiety Scale Japanese version) total score from baseline to Week 12 of the treatment period | Up to 19 weeks

SECONDARY OUTCOMES:
The transition of LSAS-J(Liebowitz Social Anxiety Scale Japanese version) total score from baseline to Week 8 of the treatment period | Up to 19 weeks
The transition of LSAS-J(Liebowitz Social Anxiety Scale Japanese version) Fear or Anxiety score from baseline to Week 8 of the treatment period | Up to 19 weeks
The transition of LSAS-J(Liebowitz Social Anxiety Scale Japanese version) Avoidance score from baseline to Week 8 of the treatment period | Up to 19 weeks
Responder rates of LSAS-J(Liebowitz Social Anxiety Scale Japanese version) total score at 1, 2, 4, 6, 8,10and 2 weeks of the treatment period | Up to 19 weeks
  Responder is defined as a reduction of 30% or more in LSAS-J(Liebowitz Social Anxiety Scale Japanese version)total score from baseline
Remitted patient rates of LSAS-J(Liebowitz Social Anxiety Scale Japanese version) total score at 1, 2, 4, 6, 8, 10 and 12 weeks of the treatment period | Up to 19 weeks
  Remitted patient is defined as a LSAS-J(Liebowitz Social Anxiety Scale Japanese version) total score of 30 or less.
Transition of CGI-S(Clinical Global Impression of illness Severity) score from baseline to Week 12 of the treatment period | Up to 19 weeks
Transition of SDISS(Sheehan Disability Scale) score from baseline to Week 12 of the treatment period | Up to 19 weeks
Plasma ONO-1110 concentrations | Up to 19 weeks
Adverse Events | Up to 19 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (27):
- Japan (27):
  - Aisakura Clinic, Fukuoka
  - AK Clinic, Fukuoka
  - Hiro Mental Clinic, Fukuoka
  - Hirota Clinic, Fukuoka
  - Kokorono Clinic Hirao, Fukuoka
  - Kokura Mental Clinic, Fukuoka
  - Mental Clinic Sakurazaka, Fukuoka
  - Shinseikai Kaku Mental Clinic, Fukuoka
  - Uematsu Mental Clinic, Fukuoka
  - Ichikawa Clinic, Gunma
  - Higashi-Sapporo Mental Clinic, Hokkaido
  - Kawamura Mental Clinic, Hokkaido
  - Minami1jo Mental Clinic, Hokkaido
  - Sapporo Kobushi Clinic, Hokkaido
  - Shimode Mental Clinic, Hokkaido
  - Tatsuta Clinic, Hyōgo
  - Yutaka Clinic, Kanagawa
  - Ai Clinic, Miyazaki
  - Inoue Clinic, Osaka
  - Yamaguchi Mental Clinic, Tokushima
  - Harai Clinic, Tokyo
  - Iidabashi Mental Clinic, Tokyo
  - Ikebukuro Olive Mental Clinic, Tokyo
  - Maynds Tower Mental Clinic, Tokyo
  - Meguroeki Higashiguchi Mental Clinic, Tokyo
  - Monzen-nakacho Mental Clinic, Tokyo
  - Sangenjaya Nakamura Mental Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: No